CLINICAL TRIAL: NCT00000148
Title: Advanced Glaucoma Intervention Study (AGIS)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NEI-49
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2006-06-05 (Estimated); Status verified 2003-10

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy

INTERVENTIONS:
Procedure: Argon Laser Trabeculoplasty
Procedure: Trabeculectomy

SUMMARY:
To assess the long-range outcomes of sequences of interventions involving trabeculectomy and argon laser trabeculoplasty in eyes that have failed initial medical treatment for glaucoma.

DETAILED DESCRIPTION:
In advanced glaucoma, medication alone no longer reduces intraocular pressure adequately, and the eye has field defects. Before 1980, some type of filtering surgery, such as trabeculectomy, was the usual method of intervention. Since then, laser trabeculoplasty has become a popular alternative. Sometimes the first intervention chosen succeeds in controlling pressure for many years; at other times, the success lasts only a few weeks or months. Because success is limited, some patients, over time, need to undergo a sequence of surgical interventions. Little is known about which sequence gives the best long-range outcome.

The Advanced Glaucoma Intervention Study (AGIS) is designed to provide a comprehensive assessment of the long-range outcomes of medical and surgical management in advanced glaucoma. The study uses visual function status to compare two intervention sequences in managing the disease.

Eligible eyes are randomly assigned to one of two intervention sequences: (1) trabeculectomy, followed by argon laser trabeculoplasty (ALT) should trabeculectomy fail, followed by a second trabeculectomy should ALT fail; or (2) ALT, followed by trabeculectomy should ALT fail, followed by another trabeculectomy should the first trabeculectomy fail. Antifibrotic agents may be used as an adjunct to trabeculectomy, but only in eyes with a previous history of invasive surgery. Eyes that fail the entire assigned sequence of interventions are managed at the discretion of the AGIS physician in collaboration with the patient.

Interventions are supplemented with medical treatment as needed. A total of 789 eyes with advanced glaucoma have been enrolled. All patients are being followed under a standardized protocol for a minimum of 5 years to determine degree of visual function loss, failure rates of interventions, rates of complications, and need for supplemental therapy.

After the initial intervention, followup examinations are scheduled at 1 week, 4 weeks, 3 months, 6 months, and every 6 months thereafter. After second and third interventions, followup examinations are scheduled at 1 and 4 weeks. Additional visits are scheduled as necessary for the management of the disease.

The primary outcome variable in AGIS is average percent of eyes with decrease of vision, where decrease of vision is a substantial decline of either visual field or visual acuity attributable to the effect of glaucoma. Secondary outcome variables include sustained decrease of vision, failure of interventions, number of prescribed glaucoma medications, and level of intraocular pressure. An ancillary study is assessing filtering bleb encapsulation.

ELIGIBILITY:
Men and women between the ages of 35 and 80 with open-angle glaucoma that was not successfully controlled by medication were eligible for enrollment.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1988-04

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Yale University School of Medicine, Yale Eye Center, New Haven, Connecticut
  - Georgetown University, University Ophthalmic Consultants of Washington, Eye Associates of Washington, D.C., Washington D.C., District of Columbia
  - Emory University, Emory Eye Center, Atlanta, Georgia
  - Piedmont Hospital, Eye Consultants of Atlanta, Atlanta, Georgia
  - Humana Health Plan Sykes Center, Chicago, Illinois
  - University of Illinois, Eye and Ear Infirmary, Chicago, Illinois
  - Washington Hospital Center, Washington Eye Physicians and Surgeons, Chevy Chase, Maryland
  - University of Michigan, W.K. Kellogg Eye Center, Ann Arbor, Michigan
  - Sinai Hospital, Detroit, Franklin Eye Consultants, Southfield, Michigan
  - Ohio State University, Department of Ophthalmology, Ophthalmic Surgeons and Consultants, Columbus, Ohio
  - Wills Eye Hospital, Glaucoma Service, Philadelphia, Pennsylvania
  - University of Virginia Medical Center, Department of Ophthalmology, Charlottesville, Virginia
  - Medical College of Virginia, Department of Ophthalmology, Richmond, Virginia

REFERENCES:
- [Background] The Advanced Glaucoma Intervention Study (AGIS) Manual of Operations. Springfield, Virginia., National Technical Information Service, 1993;No. PB93-220192
- [Background] Ederer F, Gaasterland DE, Sullivan EK; AGIS Investigators. The Advanced Glaucoma Intervention Study (AGIS): 1. Study design and methods and baseline characteristics of study patients. Control Clin Trials. 1994 Aug;15(4):299-325. doi: 10.1016/0197-2456(94)90046-9. PMID 7956270
- [Background] Advanced Glaucoma Intervention Study. 2. Visual field test scoring and reliability. Ophthalmology. 1994 Aug;101(8):1445-55. PMID 7741836
- [Background] The Advanced Glaucoma Intervention Study (AGIS) Data Management Handbook. Springfield, Virginia., National Technical Information Service, Document, 1996;No. PB96-137120
- [Background] The Advanced Glaucoma Intervention Study (AGIS): 3. Baseline characteristics of black and white patients. Ophthalmology. 1998 Jul;105(7):1137-45. doi: 10.1016/s0161-6420(98)97012-9. PMID 9663214
- [Background] The Advanced Glaucoma Intervention Study (AGIS): 4. Comparison of treatment outcomes within race. Seven-year results. Ophthalmology. 1998 Jul;105(7):1146-64. doi: 10.1016/s0161-6420(98)97013-0. PMID 9663215
- [Derived] Caprioli J, Mock D, Bitrian E, Afifi AA, Yu F, Nouri-Mahdavi K, Coleman AL. A method to measure and predict rates of regional visual field decay in glaucoma. Invest Ophthalmol Vis Sci. 2011 Jul 1;52(7):4765-73. doi: 10.1167/iovs.10-6414. PMID 21467178